CLINICAL TRIAL: NCT04401891
Title: The Benefit of Formal Pre-operative Education to Patient Satisfaction, Pain and Function
Brief Title: Formal Pre-Operative Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201911175
Record Dates: First submitted 2020-05-13; First posted 2020-05-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Upper Extremity Orthopedic Surgery Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Pre-Operative Education in MD office prior to surgery (No Intervention)
- Formal Pre-operative education/therapy prior to surgery (Experimental)
  Interventions: Behavioral: Formal pre-operative education

INTERVENTIONS:
Behavioral: Formal pre-operative education — One group of patients will receive formal pre-operative education prior to surgery from an occupational or physical therapists while the other group of patients will only receive routine education in the MD office.
  Arms: Formal Pre-operative education/therapy prior to surgery

SUMMARY:
The investigators want to determine if delivering formal preoperative education to patients helps the patients with post operative pain, function and overall satisfaction. Education would cover surgery, post operative activities of daily living, pain and edema management, duration of recovery and any expected therapy they might need. All participants will receive a pre and post operative questionnaire to determine level of understanding of anticipated needs and barriers due to surgery. Group one will receive formal education from an occupational therapist or physical therapist while Group two will receive only standard education in the MD clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* English as Primary language,
* scheduled to have orthopedic upper extremity surgery.

Exclusion Criteria:

* less than 18 years
* Conservative management or non operative management of orthopedic upper extremity surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
PROMIS (Patient-Reported Outcomes Measurement Information System) Physical Function Subtest -- change is being assessed | prior to surgery and two weeks post surgery
  Bell curve scale for scoring: A score of 50 is the average amount of physical function and/or upper extremity function in the general population. A score below 40 would be poorer function, whereas, a score above 60 would be better function than the general population.
PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety subtest -- change is being assessed | prior to surgery and two weeks post surgery
  Bell Curve scale for scoring:A score of 50 is the average amount of anxiety in the general public. A score above 60 the patient has significant anxiety
PROMIS (Patient-Reported Outcomes Measurement Information System) Depression subtest -- change is being assessed | prior to surgery and two weeks post surgery
  Bell shape curve scoring: A score of 50 is the average amount for depression in the general public. A score above 60 corresponds to a score of 10 on the Patient Health Questionnaire (PHQ)-9 scale, which is the cutoff with the highest sensitivity and specificity to detect a diagnosis of moderately severe major depression.
PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference subtest -- change is being assessed | prior to surgery and two weeks post surgery
  Bell shape curve scoring: The higher the score above 50 the more the pain the lower the score below 50 the less the pain
PROMIS (Patient-Reported Outcomes Measurement Information System)Upper Extremity Function subtest -- change is being assessed | prior to surgery and two weeks post surgery
  Bell shape curve scoring:A score of 50 is the average amount of physical function and/or upper extremity function in the general population. A score below 40 would be poorer function, whereas, a score above 60 would be better function than the general population.
MODEMS (Musculoskeletal Outcomes Data Evaluation Management Scale) Pre-Operative | prior to surgery
  1 to 5 scale with 1 being not at all likely and 5 being extremely likely. Also is a 6 for not applicable
MODEMS (Musculoskeletal Outcomes Data Evaluation Management Scale) post operative | 2 weeks post surgery
  1 to 5 scale with 1 being not at all likely and 5 being extremely likely. Also is a 6 for not applicable
Pain Scale | prior to surgery and 2 weeks post surgery
  0 to 10 likert scale. 0 being no pain and 10 being worst pain possible

CONTACTS AND LOCATIONS:
Overall Officials: Logan Berlet, OTD, Principal Investigator — Washington University in Saint Louis
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No